CLINICAL TRIAL: NCT04720599
Title: Clinical Evaluation of ExoDx™ Prostate(IntelliScore) in Men Presenting for Initial Prostate Biopsy
Brief Title: Clinical Evaluation of ExoDx Prostate(IntelliScore) in Men Presenting for Initial Prostate Biopsy
Status: Completed | Type: Observational
Sponsor: Exosome Diagnostics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ECT2020-002
Record Dates: First submitted 2021-01-20; First posted 2021-01-22 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2020-12

CONDITIONS: Urologic Cancer
Keywords: exosome; ExoDx Prostate
MeSH Terms: conditions — Urologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: ExoDx Prostate(IntelliScore) — The ExoDx Prostate test result supports the biopsy decision process by stratifying patients based on risk for high grade prostate cancer
  Other Names: EPI; EPI-CE

SUMMARY:
The study described here is being conducted to prospectively confirm the performance of the ExoDx Prostate gene expression assay in patients presenting for an initial prostate biopsy and support of CE-marking the test for a European Union Launch.

ELIGIBILITY:
Inclusion Criteria:

* Clinical suspicion for prostate cancer
* Elevated Prostate-specific Antigen between 2.0-10 ng/ mL
* Scheduled for a initial prostate biopsy

Exclusion Criteria:

* Clinical symptoms of urinary tract infection (including prostatitis) at the time of enrollment.
* History of prostate cancer.
* History of invasive treatments for benign prostatic hypertrophy (BPH) or lower urinary track symptoms within 6 months of study enrollment.
* Known hepatitis status (all types) and/or HIV documented in patient's medical record.
* Patients with history of concurrent renal/bladder tumors.
* Prior MRI used in the decision to biopsy

Min Age: 50 Years | Sex: Male
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants with prostates
Study Population: - Men, aged 50yrs or older with an elevated PSA between 2-10ng/ml scheduled for an initial biopsy
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Correlation of the ExoDx Prostate test results with the outcome of prostate biopsies in an initial biopsy patient cohort. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Mikkel Noerholm, Study Director — Exosome Diagnostics, Inc.
Locations (3):
- United States (2):
  - Chesapeake Urology Research Associates, Baltimore, Maryland
  - New Jersey Urology, Voorhees Township, New Jersey
- Klinikum der Universität München, München, Germany

IPD SHARING:
Plan to Share IPD: Yes
IPD can be shared on an individual basis. Please reach out for more information.
Supporting Information: Study Protocol, ICF
Time Frame: 12 months after trial completion
Access Criteria: Individual basis upon mutual agreement

REFERENCES:
- [Derived] Kretschmer A, Kajau H, Margolis E, Tutrone R, Grimm T, Trottmann M, Stief C, Stoll G, Fischer CA, Flinspach C, Albrecht A, Meyer L, Priewasser T, Enderle D, Muller R, Torkler P, Alter J, Skog J, Noerholm M. Validation of a CE-IVD, urine exosomal RNA expression assay for risk assessment of prostate cancer prior to biopsy. Sci Rep. 2022 Mar 21;12(1):4777. doi: 10.1038/s41598-022-08608-z. PMID 35314720
- [Derived] Kretschmer A, Tutrone R, Alter J, Berg E, Fischer C, Kumar S, Torkler P, Tadigotla V, Donovan M, Sant G, Skog J, Noerholm M. Pre-diagnosis urine exosomal RNA (ExoDx EPI score) is associated with post-prostatectomy pathology outcome. World J Urol. 2022 Apr;40(4):983-989. doi: 10.1007/s00345-022-03937-0. Epub 2022 Jan 27. PMID 35084544